CLINICAL TRIAL: NCT03945305
Title: Safety and Efficacy of Remote Ischemic Conditioning Treatment for Community-based Essential Hypertension: a Randomized, Parallel-controlled Clinical Trial
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning Treatment for Community-based Essential Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SERIC-EH
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension, Remote Ischemic Conditioning
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): Patients are treated with previous antihypertensive treatment plus remote ischemic conditioning.
  Interventions: Device: Patients are treated with previous antihypertensive treatment plus remote ischemic conditioning.
- Control group (Other): Patients are only treated with previous antihypertensive treatment.
  Interventions: Other: Previous antihypertensive treatment

INTERVENTIONS:
Device: Patients are treated with previous antihypertensive treatment plus remote ischemic conditioning. — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg.
  Arms: RIC group
Other: Previous antihypertensive treatment — Patients are only treated with previous antihypertensive treatment.
  Arms: Control group

SUMMARY:
The purpose of this study is to explore the efficacy and safety of remote ischemic conditioning for essential hypertension in the community population.

DETAILED DESCRIPTION:
At present, stroke has become the leading cause of death in China, with hypertension being the primary risk factor and one of the controllable risk factors. Current studies have shown that remote ischemic conditioning can improve vascular endothelial function, inhibit sympathetic nervous system activity and regulate immune and inflammatory reactions. Thus it may exert anti-hypertensive effects through multiple mechanisms. The purpose of this study is to investigate the efficacy and safety of remote ischemic conditioning for essential hypertension in the community population.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥40 years, ≤ 75 years, regardless of sex;
2. Having the history of essential hypertension and the systolic blood pressure of at least 140 mm Hg on two consective days;
3. Signed and dated informed consent is obtained

Exclusion Criteria:

1. Blood pressure ≥ 180/110mmHg;
2. Planned adjustment of antihypertensive drugs in the next month;
3. Severe hematologic disorders or significant coagulation abnormalities;
4. Individuals who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper limb, acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
5. Pregnant or lactating women;
6. Severe hepatic and renal dysfunction, or ALT/AST >3 times upper limit of normal, or serum creatinine >265umol/l (>3mg/dl);
7. Patients being enrolled or having been enrolled in another clinical trial within the 3 months prior to this clinical trial;
8. Patients unsuitable for enrollment in the clinical trial according to the investigator's discretion.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Changes of mean systolic blood pressure | 12-14 days
  The mean systolic blood pressure in the last 3 days of treatment minus baseline mean systolic blood pressure

SECONDARY OUTCOMES:
Mean systolic blood pressure level | 12-14 days
  Mean systolic blood pressure levels during the last 3 days of treatment
Changes of mean diastolic blood pressure | 12-14 days
  The mean diastolic blood pressure in the last 3 days of treatment minus baseline mean diastolic blood pressure
Mean diastolic blood pressure level | 12-14 days
  Mean diastolic blood pressure levels during the last 3 days of treatment
Blood pressure compliance rate | 15-28 days
  Blood pressure compliance rates after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China